CLINICAL TRIAL: NCT07294170
Title: A Master Protocol for an Exploratory, Phase 2a, Proof-of-Concept Platform Study to Evaluate the Safety, Tolerability, and Efficacy of Multiple Regimens in Participants With Myasthenia Gravis
Brief Title: ADAPT Forward - Master Protocol of a Platform Study to Evaluate the Safety and Efficacy of Multiple Regimens in Participants With Myasthenia Gravis
Status: Recruiting | Type: Observational
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Other Study IDs: ARGX-999-2-MG-2000
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Myasthenia Gravis; MG; gMG; Generalized Myasthenia Gravis; Generalized Myasthenia Gravis (gMG); AChR-Ab Seropositive Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ISA1 participants: Participants With AChR-Ab Seropositive Generalized Myasthenia Gravis With a Partial Clinical Response to Efgartigimod
  Interventions: Biological: Efgartigimod IV; Biological: Empasiprubart IV

INTERVENTIONS:
Biological: Efgartigimod IV — Intravenous infusion of efgartigimod
Biological: Empasiprubart IV — Intravenous infusion of empasiprubart

SUMMARY:
ADAPT Forward is a platform study with the aim to look at how safe different drugs are and how well they work for people with myasthenia gravis. The goal is to find the best therapeutic approach to reduce patients' side effects and improve their quality of life.

DETAILED DESCRIPTION:
This is a platform study and is governed by a single master protocol that enables multiple regimens to be evaluated in separate intervention-specific appendixes (ISAs).

The key design structure of the platform study comprises: common master protocol screening period, ISA-specific screening period, ISA treatment period of variable duration and design and ISA safety follow-up/follow-up period of variable duration.

Details on each study period will be specified in the ISAs. Following ISAs are included in this platform study:

* NCT07284420 - ADAPT Forward 1 - a study to evaluate empasiprubart IV as add-on therapy to efgartigimod IV in participants with AChR-Ab seropositive generalized myasthenia gravis with a partial clinical response to efgartigimod (https://www.clinicaltrials.gov/study/NCT07284420)

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and the local legal age of consent for clinical studies
* Has been diagnosed with MG with consistent clinical features per the investigator's clinical judgment
* If receiving MG therapy, including nonsteroidal immunosuppressive drugs (NSIDs), corticosteroids, or acetylcholinesterase (AChE) inhibitors either in combination or alone, the participant should receive a stable dosage before master protocol screening

Exclusion Criteria:

* Known autoimmune disease or any medical condition other than the indication under study that would interfere with an accurate assessment of clinical symptoms of MG or puts the participant at undue risk
* Is MGFA (Myasthenia Gravis Foundation of America) Class V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants With AChR-Ab Seropositive Generalized Myasthenia Gravis With a Partial Clinical Response to Efgartigimod
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2028-03-07 (Estimated); Study Completion 2028-03-07 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of multiple regimens (monotherapy or add-on therapy to backbone therapy) in MG subtypes | Up to approximately 7 years (the duration of each ISA will vary and be specified on the ISA records)

SECONDARY OUTCOMES:
To evaluate the efficacy of multiple regimens (monotherapy or add-on therapy to backbone therapy) in MG subtypes | Up to approximately 7 years (the duration of each ISA will vary and be specified on the ISA records)
  Each ISA record will specify the correct scale and time point

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Profound Research LLC - Carlsbad, Carlsbad, California
  - Visionary Investigators Network, Miami, Florida
  - National Neuromuscular Research Institute, Austin, Texas

IPD SHARING:
Plan to Share IPD: No